CLINICAL TRIAL: NCT00251199
Title: A Phase 1b Viral Kinetic Study of VX-950 and Peginterferon in Hepatitis C
Brief Title: VX-950 and Peginterferon for Hepatitis C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: VX05-950-103
Record Dates: First submitted 2005-11-07; First posted 2005-11-09 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir

INTERVENTIONS:
Drug: VX-950
Drug: peginterferon

SUMMARY:
VX-950 is an investigational drug , which is being tested in combination with a known treatment for hepatitis C, peginterferon.

ELIGIBILITY:
Inclusion Criteria:

* infected with Hepatitis C virus

Exclusion Criteria:

* contraindications to peginterferon therapy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Enrollment: 20
Dates: Start 2005-10; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Viral kinetics

SECONDARY OUTCOMES:
Assess the safety of VX-950 in combination with peginterferon

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (2):
- Call for information, Homburg/Saar, Germany
- Call for information, Amsterdam, Netherlands